CLINICAL TRIAL: NCT06998095
Title: Tezepelumab (Tezspire) Regulatory Postmarketing Surveillance in Korea
Acronym: Tezepelumab
Status: Not yet recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5180R00020
Record Dates: First submitted 2025-05-29; First posted 2025-05-31 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Severe Asthma
Keywords: severe asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The objectives of this study are to describe the occurrence of adverse events and the effectiveness of tezepelumab in patients receiving tezepelumab as indicated for severe asthma in South Korea.

DETAILED DESCRIPTION:
Primary objective(s):

* To estimate the incidence proportion of adverse events (AEs), adverse drug reactions (ADR1s), serious adverse events (SAEs), serious adverse drug reaction (SADRs), unexpected2 adverse events, unexpected adverse drug reactions and expected adverse drug reactions, separately among patients receiving tezepelumab for severe asthma in routine clinical practice.
* To describe the nature (type), severity, and causality of adverse events (AEs)/adverse drug reactions (ADRs) and actions taken to address AEs among patients receiving tezepelumab for severe asthma in routine clinical practice.

Secondary objective(s) :

* To estimate the proportion of patients with improved asthma control from baseline to week 24 after tezepelumab initiation or the last known routine visit [i.e., end of treatment (EoT)]
* To estimate the incidence rate of adverse events (AEs) , adverse drug reactions (ADRs), serious adverse events (SAEs), serious adverse drug reaction (SADRs), unexpected adverse events, unexpected adverse drug reactions and expected adverse drug reactions per unit time, separately among patients receiving tezepelumab for severe asthma in routine clinical practice.

Exploratory Objective(s):

* To estimate the incidence proportion of AEs by demographic and clinical characteristics
* To estimate the proportion of patients with improved asthma control from baseline to week 24 after tezepelumab initiation or the last known routine visit by demographic and clinical characteristics

This is a prospective, single-arm, multicenter, observational study to evaluate the safety and effectiveness of tezepelumab from treatment initiation up to 24 weeks in patients who are prescribed tezepelumab according to its approved indication for severe asthma in South Korea.

The asthma control effectiveness assessment will be an evaluation of change from treatment initiation up to 24 weeks after treatment initiation. This study design will reflect the actual management of these subjects in routine clinical practice. The treating physician will determine the treatment plan, as well as the frequency of laboratory and clinical assessment, if necessary, based on routine practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are treated with at least one dose of tezepelumab according to the indication in the locally approved prescribing information
2. Patients with evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study

Exclusion Criteria:

1. Other off-label indications according to the locally approved prescribing information
2. Current participation in any interventional trial

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study Population:
  The study population will consist of adolescent and adult patients with a diagnosis of severe asthma who are receiving tezepelumab according to its approved indication by MFDS. Eligible patients will be enrolled by a continuous registration method.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-11-28 (Estimated); Primary Completion 2029-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events (AEs), adverse drug reactions (ADRs), serious AEs (SAEs), serious ADRs (SADRs), unexpected AEs/ADRs, unexpected SAEs/SADRs) | up to 24 weeks
  To estimate the incidence proportion of adverse events (AEs), adverse drug reactions (ADRs), serious adverse events (SAEs), serious adverse drug reaction(SADRs), unexpected adverse events, unexpected adverse drug reactions and expected adverse drug reactions, separately among patients receiving tezepelumab for severe asthma in routine clinical practice.
  To describe the nature (type), severity, and causality of adverse events (AEs)/adverse drug reactions (ADRs) and actions taken to address AEs among patients receiving tezepelumab for severe asthma in routine clinical practice.

SECONDARY OUTCOMES:
A measure of asthma control at week 24 or at the last known routine visit as assessed by study investigator according to GINA guidelines | up to 24 weeks
  -To estimate the proportion of patients with improved asthma control from baseline to week 24 after tezepelumab initiation or the last known routine visit [i.e., end of treatment (EoT)]
Safety (adverse events (AEs), adverse drug reactions (ADRs), serious AEs (SAEs), serious ADRs (SADRs), unexpected AEs/ADRs, unexpected SAEs/SADRs) | up tp 24 weeks
  To estimate the incidence rate of adverse events (AEs) , adverse drug reactions (ADRs), serious adverse events (SAEs),serious adverse drug reaction (SADRs), unexpected adverse events, unexpected adverse drug reactions and expected adverse drug reactions per unit time, separately among patients receiving tezepelumab for severe asthma in routine clinical practice.

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/